CLINICAL TRIAL: NCT02374385
Title: A Phase 1 Randomized, Single-Center, Double-Blind, Placebo Controlled, Dose-Ranging Study to Evaluate the Safety and Immunogenicity of the BPSC-1001 (VSVΔG-ZEBOV) Ebola Virus Vaccine Candidate in Healthy Adult Subjects
Brief Title: Phase I Trial to Assess the Safety, Tolerability and Immunogenicity of a Ebola Virus Vaccine
Acronym: VSVΔG-ZEBOV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); NewLink Genetics Corporation (Industry)
Responsible Party: Principal Investigator, Scott Halperin, Dr. Scott Halperin, Dalhousie University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CI1401
Record Dates: First submitted 2015-01-06; First posted 2015-02-27 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Ebola Viruses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 1x10(5) pfu VSV G-ZEBOV vaccine (BPSC1001) each dose, total volume 1 mL
  Interventions: Biological: BPSC-1001 (VSVΔG-ZEBOV)
- Group 2 (Experimental): 5x10(5) pfu VSV G-ZEBOV vaccine (BPSC1001) each dose, total volume 1 mL
  Interventions: Biological: BPSC-1001 (VSVΔG-ZEBOV)
- Group 3 (Experimental): 3x10(6) pfu VSV G-ZEBOV vaccine (BPSC1001) each dose, total volume 1 mL.
  Interventions: Biological: BPSC-1001 (VSVΔG-ZEBOV)
- Group 4 (Placebo Comparator): Group 4 will receive placebo (normal saline).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BPSC-1001 (VSVΔG-ZEBOV) — Ebola vaccine candidate
  Other Names: BPSC-1001
  Arms: Group 1; Group 2; Group 3
Other: Placebo — Normal saline
  Arms: Group 4

SUMMARY:
Background:

Ebola virus has infected and killed people, mostly in Africa. In 2014, the Ebola virus has affected several thousand people. There is no approved effective way to treat or prevent Ebola. Researchers are trying to develop a vaccine for it.

Objectives:

To study the anti-Ebola vaccine VSV ZEBOV (BPSC1001) to see if it is safe. Also, to see how it affects people's immune system.

Eligibility:

- Healthy men and women ages 18-65. They must not have a chronic medical condition that requires medicine. They must not be a healthcare worker, an animal care worker, or a childcare worker, and they must not have a household contact that has a compromised immune system, is pregnant, or is under the age of 5 years.

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Participants will be randomly assigned to get the vaccine or the placebo.
* At visit 1 (vaccination), vital signs will be taken and blood will be drawn. The vaccine or placebo will be injected into the upper arm muscle.
* Participants will return to the clinic 11 times over the next 6 months. Participants will have blood drawn at every study visit. Their mouth will be swabbed and urine tested at least four times after vaccination.
* For 14 days after vaccination, participants will write down their temperature, any symptoms, and any redness at the injection site. They will bring the booklet to each study visit.

All visits take place at the Canadian Center for Vaccinology, Dalhousie University/IWK Health Centre, Halifax, NS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or non-pregnant, non-lactating female, ages 18 to 65 (inclusive) at the time of screening
* Have provided written informed consent before screening
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination prior to entry into the study
* Available, able, and willing to participate for all study visits and procedures
* Males and females who are willing to practice abstinence from sexual intercourse, or are willing to use effective methods of contraception, from at least 30 days prior to vaccination until study end.

  * If the female partner is NOT of childbearing potential, the couple will only be required to use condoms, without other adjunctive contraception.
  * For this study, a woman is considered of childbearing potential unless postmenopausal (≥ 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  * Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example:
  * Male condoms PLUS: Oral contraceptives, either combined or progestogen alone, injectable progestogen,implants of etonogestrel or levonorgestrel, oestrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device or intrauterine system
* Be willing to minimize blood and body fluid exposure of others for 7 days after vaccination

  * Use of effective barrier prophylaxis, such as latex condoms, during penetrative sexual intercourse
  * Avoiding the sharing of needles, razors, or toothbrushes
  * Avoiding open-mouth kissing

Exclusion Criteria:

* History of prior infection with a filovirus or prior participation in a filovirus vaccine trial
* History of prior infection with VSV or receipt of a VSV vectored vaccine
* Is a healthcare worker who has direct contact with patients
* Has a house-hold contact (HHC) who is immunodeficient, HIV-positive, pregnant, has an unstable medical condition, or is under the age of 5 years
* Is a childcare worker who has direct contact with children 5 years of age or younger
* Directly prepares food in the food industry
* History of employment in an industry involved in contact with ruminant animals, veterinary sciences, or other potential exposure to VSV
* History of employment or activity which involves potential contact with filoviruses
* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
* Known allergy to the components of the BPSC-1001 vaccine product
* Receipt of investigational product up to 30 days prior to enrollment or ongoing participation in another clinical trial involving an investigational product
* Receipt of licensed vaccines within 30 days of planned study immunization
* Ability to observe possible local reactions at the eligible injections sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
* Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, ECG, and/or laboratory screening test
* Any baseline laboratory screening tests which is outside of acceptable range as defined in the protocol ALT, AST, creatinine, hemoglobin, platelet count, total white blood cell count, urine protein, urine occult blood, urine glucose
* Any serologic evidence of hepatitis B or C infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, cytotoxic therapy in the previous 5 years, and/or diabetes
* Any chronic or active neurologic disorder, including migraines, seizures, and epilepsy, excluding a single febrile seizure as a child
* Have an active malignancy or history of metastatic or hematologic malignancy
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years
* Moderate or severe illness and/or fever greater than 100.4 F within one week prior to vaccination
* Pregnant or lactating female, or female who intends to become pregnant during the study period
* Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
* History of blood donation within 60 days of enrollment or plans to donate within the study period
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of study entry

  * For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
  * Intranasal and topical steroids are allowed
* Unwilling to allow storage and use of blood for future vaccine research
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local injection site reactogenicity signs and symptoms: pain, erythema, and induration | 2 months
Frequency of adverse events (AEs), severity and assessed relationship to study products | 2 months
Distribution of values of safety laboratory measures at baseline and at follow-up visits post-vaccination | 3 months
Number of participants with early discontinuation of vaccinations and reason for discontinuation | 3 months

SECONDARY OUTCOMES:
Measurement of ZEBOV envelope glycoprotein-specific binding antibody by ELISA | 6 months
rVSV in blood, urine, or saliva as detected by real-time polymerase chain reaction [RT-PCR] | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Halperin, MD, Principal Investigator — Dalhousie University

REFERENCES:
- [Derived] Coller BG, Blue J, Das R, Dubey S, Finelli L, Gupta S, Helmond F, Grant-Klein RJ, Liu K, Simon J, Troth S, VanRheenen S, Waterbury J, Wivel A, Wolf J, Heppner DG, Kemp T, Nichols R, Monath TP. Clinical development of a recombinant Ebola vaccine in the midst of an unprecedented epidemic. Vaccine. 2017 Aug 16;35(35 Pt A):4465-4469. doi: 10.1016/j.vaccine.2017.05.097. Epub 2017 Jun 21. PMID 28647166
- [Derived] ElSherif MS, Brown C, MacKinnon-Cameron D, Li L, Racine T, Alimonti J, Rudge TL, Sabourin C, Silvera P, Hooper JW, Kwilas SA, Kilgore N, Badorrek C, Ramsey WJ, Heppner DG, Kemp T, Monath TP, Nowak T, McNeil SA, Langley JM, Halperin SA; Canadian Immunization Research Network. Assessing the safety and immunogenicity of recombinant vesicular stomatitis virus Ebola vaccine in healthy adults: a randomized clinical trial. CMAJ. 2017 Jun 19;189(24):E819-E827. doi: 10.1503/cmaj.170074. PMID 28630358